CLINICAL TRIAL: NCT03383185
Title: Metabolic Profile of Users of Hormonal and Non-hormonal Contraceptives, 5-year Follow-up
Brief Title: Metabolic Profile of Users of Hormonal and Non-hormonal Contraceptives
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, PhD, Federal University of São Paulo
Other Study IDs: CAAE: 45523715.4.0000.5505
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Contraceptive Usage; Metabolic Syndrome; Body Weight Changes
Keywords: contraception; Body mass index; Metabolic Syndrome; obesity
MeSH Terms: conditions — Contraception Behavior; Metabolic Syndrome; Body Weight Changes; Obesity | interventions — Intrauterine Devices; Contraceptives, Oral, Combined; Medroxyprogesterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-hormonal contraceptive: Users of non- hormonal intrauterine device during the 5 years follow-up
  Interventions: Device: Intrauterine device
- Hormonal contraceptives: Users of combined oral contraceptive, progestin-only pills, depot-medroxyprogestereone acetate during 5 years follow-up
  Interventions: Drug: Combined Oral Contraceptive; Drug: Progestin-only pills; Drug: Depot-Medroxyprogestereone Acetate

INTERVENTIONS:
Device: Intrauterine device — Use of Intrauterine device during the follow-up period
  Groups: Non-hormonal contraceptive
Drug: Combined Oral Contraceptive — Use of combined oral contraceptive during the follow-up period
  Groups: Hormonal contraceptives
Drug: Progestin-only pills — Use of progestin-only pills during the follow-up period
  Groups: Hormonal contraceptives
Drug: Depot-Medroxyprogestereone Acetate — Use of depot-medroxyprogesterone acetato during the follow-up period
  Groups: Hormonal contraceptives

SUMMARY:
Evaluation of metabolic profile of users of hormonal and non-hormonal contraceptives during five years follow-up

DETAILED DESCRIPTION:
Were eligible for the study 489 Women, followed in Federal University of São Paulo Family Planning Service, who used the same contraceptive method during five year of follow-up, According to the service protocol, the patients, after had participated of a orientation group about contraceptives methods, elected one of them. After that, if the choice had been according to the eligibility criteria of World Health Organization, it was approved by a gynecologist.

The contraceptive methods available were the intrauterine device (IUD) oral contraceptives, including combined pills and progestin-only formulations, and depot medroxyprogestereone acetate.

The study consisted in the evaluation of their medical records of weight, BMI, Blood pressure, glycemia, seric levels of cholesterol and triglycerides, during the five years, and in the comparison of the differences of these data between the contraceptive methods.

ELIGIBILITY:
Inclusion Criteria:

* women in reproductive age followed in Federal university of Sao Paulo Family Planning Service
* use of the same contraceptive method during five years

Exclusion Criteria:

* incomplete data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women in menacme, users of the same contraceptive hormonal (combined oral contraceptives, progestin-only pills and depot-medroxyprodestereone acetate) and non-hormonal contraceptive methods (IUD) during five years
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | five years follow-up
  evaluation of variation of body mass index during the usage of hormonal and non-hormonal contraceptives

SECONDARY OUTCOMES:
glycemia | five years follow-up
  evaluation of variation of glycemia during the usage of hormonal and non-hormonal contraceptives
cholesterol level | five years follow-up
  evaluation of variation of cholesterol serum levels during the usage of hormonal and non-hormonal contraceptives
triglycerides level | five years follow-up
  evaluation of variation of triglycerides serum levels during the usage of hormonal and non-hormonal contraceptives

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo - Unifesp, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided